CLINICAL TRIAL: NCT04061902
Title: Participation in Surgical Cancer Care; Patient, Next of Kin and Health Care Professionals' Perspective
Brief Title: Participation in Surgical Cancer Care
Acronym: Particip
Status: Completed | Type: Observational
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Jenny Drott, Registered nurse, PhD, Ostergotland County Council, Sweden
Other Study IDs: Part.19
Record Dates: First submitted 2019-08-16; First posted 2019-08-20 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Participation with enhanced patient perioperative information — Improved information and dialogue about the care goals in the fast track protocol.

SUMMARY:
Patients that are involved in their health care is associated with improved treatment outcomes, rehabilitation and recovery. In this research project we aim to assess patient participation among patients who had surgery for liver, bile duct (cholangiocarcinoma) and pancreatic cancer and follow a fast-track recovery program.

DETAILED DESCRIPTION:
Implementation of Fast-track surgery programs for patients with tumors in the upper GI-tract are steadily increasing because of the decreased costs, shorter hospital stays and a decrease in morbidity, mortality and post-operative complications associated with Fast-track programs. The health care team follows a standardized care program consisting of a check list with day-to-day evidence based procedures which reduces postoperative complications. Postoperative recovery is described as a process in which patients strive for a return to a normalized daily life.

Major surgeries are associated with pain, nausea, postoperative ileus , fatigue, post-operative complications such as wound infections , heart or lung dysfunctions and thromboembolic complications. In the last 20 years perioperative care, anesthesia and surgery for patients suffering from tumors has developed greatly. This has led to development and evaluation of concepts to enhance the patients recovery after different types of surgery. Fast-track surgery concepts results in decreased morbidity and enhanced recovery by implemented evidence based principles in analgesia, anesthesia, fluid management, nutrition, ambulation, minimal invasive surgery and reduction of surgical stress.

In recent years there's been a shift in focus of patient care. Patients are moving from a passive role to being more participant in their care. In Sweden, patients have the legal right to participate in their own care, and health care should be individualized for each patient's needs and abilities. Being involved in your own health care contributes to increased motivation and an improvement of the situation. This may in some cases lead to better treatment outcomes and greater satisfaction with the given care. A severe symptom burden can make the patient a passive recipient of health care without initiative or strength to be involved in the care. In patients with malignancies of the upper gastrointestinal tract monitoring and symptom relief of importance to stimulate opportunities for participation.

Aim

To investigate and describe patient participation among patients who had surgery for liver, bile duct (cholangiocarcinoma) and pancreatic cancer and follow a fast-track recovery program.

Specific aims

* To identify and describe patient participation in patients who follow a fast track-care concept
* To explore patients experiences of patient participation
* To identify, describe and evaluate patient assessed health related quality of life; and relations with patient participation

ELIGIBILITY:
Consecutive sampling strategy, patients will be screened and asked for participation both in verbal and written information. The responsibility health care professionals judge about the patient's condition to participate in the study, according to the inclusion and exclusion criteria.

Inclusion Criteria:

- patients who had surgery for liver, bile duct and pancreatic cancer and follow a fast-track recovery program >18 years old

Exclusion Criteria:

* cognitive dysfunction
* could not master the Swedish language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had surgery for liver, bile duct and pancreatic cancer and follow a fast-track recovery program.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2020-02-19 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Treatment planning | Two weeks post discharge
  Higher clinical significant score in the subscale Treatment planning in a questionnarie to measure patient participation (Arnetz et al). All scale items ask the patient to rate a specific statement on a 4-point Likert scale ranging from 1 (no, not at all) to 4 (yes, to a great degree). For all scales, higher scores indicate more positive ratings.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, County Council of Östergötland, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Amin A, Norden M, Fomichov V, Bjornsson B, Lindhoff Larsson A, Sandstrom P, Drott J. Patient-reported participation in hepatopancreatobiliary surgery cancer care: A pilot intervention study with patient-owned fast-track protocols. Eur J Cancer Care (Engl). 2022 May;31(3):e13570. doi: 10.1111/ecc.13570. Epub 2022 Mar 10. PMID 35274386